CLINICAL TRIAL: NCT07352046
Title: Effects of a Mindfulness-Based Intervention on Stress, Psychological Resilience, and Academic Self-Efficacy Among Nursing Students in Somalia: A Randomized Controlled Trial
Brief Title: Mindfulness-Based Intervention for Nursing Students in Somalia
Acronym: SOM-MIND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Fadime Koyuncu, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOM-MF-2026
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Stress; Psychological Resilience; Self Efficacy
Keywords: Mindfullnes; Nursing Students; Randomized Controlled Trial; Mental Well-Being; Somalia
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Intervention Group (Experimental): Participants receive a three-week mindfulness-based intervention delivered through weekly online sessions.
  Interventions: Behavioral: Mindfulness-Based Awareness Program
- Control group (No Intervention): Participants receive no intervention during the study period and complete baseline and post-intervention assessments only.

INTERVENTIONS:
Behavioral: Mindfulness-Based Awareness Program — The intervention consists of a three-week mindfulness-based program delivered through weekly online sessions lasting 45-60 minutes. The program includes theoretical information and guided practices focusing on mindfulness awareness, breathing awareness, and emotional awareness. Audio-recorded mindfulness exercises prepared by the researcher are shared weekly with participants via a messaging application. Participants are encouraged to practice the exercises individually in a quiet environment during the intervention period.
  Arms: Mindfulness-Based Intervention Group

SUMMARY:
This study aims to evaluate the effectiveness of a mindfulness-based intervention on stress levels, psychological resilience, and academic self-efficacy among nursing students in Somalia. Nursing students often experience high levels of stress due to academic demands, clinical training, and challenging social and environmental conditions. Mindfulness-based interventions have been shown to improve mental well-being and coping skills in various student populations, but evidence from low-resource and conflict-affected settings remains limited.

In this randomized controlled trial, nursing students will be assigned either to a mindfulness-based intervention group or to a control group receiving no intervention during the study period. The intervention consists of structured mindfulness sessions focusing on breathing awareness, body awareness, emotional regulation, and present-moment attention over a three-week period.

Outcomes including perceived stress, psychological resilience, and academic self-efficacy will be measured before and after the intervention using validated self-report instruments. The findings of this study are expected to contribute to the understanding of non-pharmacological, low-cost mental health interventions for nursing students in low-resource settings.

DETAILED DESCRIPTION:
This randomized controlled trial was designed to investigate the effects of a mindfulness-based intervention on stress, psychological resilience, and academic self-efficacy among nursing students in Somalia. Nursing students represent a population at increased risk for psychological distress due to intensive academic workloads, exposure to clinical environments, and limited mental health support resources, particularly in low-income and post-conflict settings.

The study was conducted among nursing students enrolled at a university-affiliated training institution in Mogadishu, Somalia. Eligible participants were nursing students who voluntarily agreed to participate and provided informed consent. Participants were randomly assigned to either an intervention group or a control group. The intervention group received a structured mindfulness-based program delivered over three weeks, while the control group continued with their routine academic activities without any additional intervention during the study period.

The mindfulness-based intervention included guided practices such as mindful breathing, body scan exercises, awareness of thoughts and emotions, and techniques aimed at enhancing present-moment awareness and emotional regulation. Sessions were conducted in a group format and adapted to the cultural and educational context of the participants.

Primary outcome measures included perceived stress, psychological resilience, and academic self-efficacy. These outcomes were assessed using validated questionnaires administered at baseline and after completion of the intervention. Data were analyzed to compare changes in outcome measures between the intervention and control groups.

This study seeks to provide evidence on the feasibility and effectiveness of mindfulness-based interventions as a low-cost, non-pharmacological strategy to support mental well-being and academic functioning among nursing students in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Being a nursing student enrolled in the 3rd or 4th year
* Aged 18 years or older
* Volunteering to participate in the study
* Ability to attend online sessions
* Ability to complete self-report questionnaires

Exclusion Criteria:

* Having a diagnosed psychiatric disorder
* Currently receiving psychological or psychiatric treatment
* Participation in another mindfulness or stress management program during the study period
* Inability to complete the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress Level | Baseline and 3 weeks
  Perceived stress will be assessed using the Perceived Stress Scale (PSS). The scale consists of two sub-dimensions: perceived inadequate self-efficacy and perceived stress, each originally comprising seven items. Items are rated on a 5-point Likert-type scale ranging from 0 ("Never") to 5 ("Very often"), with higher scores indicating higher perceived stress levels. Several items are reverse-coded.

SECONDARY OUTCOMES:
Change in Psychological Resilience | Baseline and 3 weeks
  Psychological resilience will be measured using the Connor-Davidson Resilience Scale - Short Form (CD-RISC-10). The scale includes 10 items rated on a 5-point Likert scale (0 = "Not true at all" to 4 = "True nearly all the time"). Higher scores reflect greater psychological resilience. The Turkish adaptation has been shown to be valid and reliable.
Change in Academic Self-Efficacy | Baseline and 3 weeks
  Academic self-efficacy will be assessed using the Academic Self-Efficacy Scale. The scale has a single-factor structure and consists of 7 items rated on a 4-point Likert-type scale, ranging from 1 ("Completely applies to me") to 4 ("Does not apply to me at all"). Total scores range from 7 to 28, with higher scores indicating higher levels of academic self-efficacy.
  The original version of the scale developed by Jerusalem and Schwarzer demonstrated good internal consistency (Cronbach's alpha = 0.87). The Turkish adaptation by Yılmaz, Gürçay, and Ekici also showed acceptable internal consistency reliability (Cronbach's alpha = 0.79).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39972317/